CLINICAL TRIAL: NCT07040020
Title: Water-Assisted Versus Standard ESD for Large Nonpedunculated Colorectal Polyps: a Prospective Randomized Trial
Brief Title: This Randomized, Single-center Trial Aims to Evaluate the Advantages of Underwater ESD (U-ESD) in Comparison to the Conventional ESD (C-ESD).
Acronym: Wave-ESD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, MD, Istituto Clinico Humanitas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID 4139 Wave-ESD
Record Dates: First submitted 2024-09-12; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Precancerous Lesions
Keywords: esd; large nonpedunculated colorectal polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional ESD (Active Comparator): Conventional ESD (C-ESD): under CO2 insufflation, initial submucosal injection of saline and methylene blue is performed; subsequent mucosal incision with ESD knife all around the lesion and submucosal dissection deep in the submucosal layer leading to an en bloc resection is carried out
  Interventions: Other: Conventional ESD (C-ESD)
- Underwater ESD (U-ESD) (Experimental): Underwater ESD (U-ESD): after filling the lumen with saline and sucking all the air, initial submucosal injection of saline and methylene blue is performed; subsequent mucosal incision with ESD knife all around the lesion and submucosal dissection deep in the submucosal layer leading to an en bloc resection is carried out.
  Interventions: Procedure: Underwater ESD (U-ESD)

INTERVENTIONS:
Procedure: Underwater ESD (U-ESD) — Underwater ESD (U-ESD): after filling the lumen with saline and sucking all the air, initial submucosal injection of saline and methylene blue is performed; subsequent mucosal incision with ESD knife all around the lesion and submucosal dissection deep in the submucosal layer leading to an en bloc resection is carried out
  Arms: Underwater ESD (U-ESD)
Other: Conventional ESD (C-ESD) — Conventional ESD (C-ESD): under CO2 insufflation, initial submucosal injection of saline and methylene blue is performed; subsequent mucosal incision with ESD knife all around the lesion and submucosal dissection deep in the submucosal layer leading to an en bloc resection is carried out.
  Arms: Conventional ESD

SUMMARY:
Large nonpedunculated colorectal lesions are increasingly detected thanks to screening programs worldwide. ESD is the technique which provides a high-quality resection of these large polyps.

Nevertheless, colorectal ESD is burdened by technical difficulties and several adverse events affecting its outcomes. The adverse events could be life-threatening, call for or prolong the hospitalization, require blood transfusion, additional endoscopic or surgical procedures and increase costs. Failure of endoscopic resection requiring surgery for benign lesions could affect patients' quality of life and increase healthcare systems' costs.

Thus, improving colorectal ESD outcomes is an important clinical and medico-economic objective. The underwater setting with saline has been already established as a better option than conventional CO2 insufflation for EMR of large colonic polyps. Moreover, use of the underwater approach for colorectal ESD has been increasingly reported with good results in the last few years. However, a randomized comparative trial between conventional and underwater colorectal ESD clarifying which should be the preferred approach is lacking.

Expected benefits are a decrease of adverse events and an increase of successful R0 resection rate of colorectal ESD.

DETAILED DESCRIPTION:
The procedure in this study involves the application of underwater ESD for the resection of large nonpedunculated colorectal polyps.

Underwater ESD is a technique wherein the polyp is removed in an en bloc fashion. The procedure initiates with the identification and delineation of the polyp borders through careful endoscopic examination. Subsequently, after filling the lumen with saline and sucking all the air, initial submucosal injection of saline and methylene blue is performed to lift the lesion. After that, subsequent mucosal incision with ESD knife all around the lesion and submucosal dissection deep in the submucosal layer leading to an en bloc resection will be performed.

The clinical practice and technique of underwater ESD and conventional ESD performed during the course of the trial, will not be modified from standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* all patients ≥ 18 years of age with indication of ESD for large (>20mm) nonpedunculated colorectal polyps
* patients who were able to give informed written consent

Exclusion Criteria:

* Suspicion of deep submucosal cancer by analysis of pit pattern (KUDO Vn)
* Suspicion of serrated/hyperplastic polyps by analysis of pit pattern (Kudo IIo)
* Polyp involving the appendix deeply (type 2 or 3 according to Toyonaga classification)
* Polyp involving the anal verge
* Polyp inside the ileo-cecal valvula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
R0 resection | 24 hours
  Rate of successful and safe endoscopic resection defined as an R0 resection with no major adverse events (defined as any major procedure-related complication, such as delayed bleeding, intraprocedural and delayed perforation or post-electrocoagulation syndrome)

SECONDARY OUTCOMES:
Compare | at 24 hours
  Compare the:
  * mean procedural time;
  * rate of en bloc resection;
  * rate of R0 resection;
  * rate of curative resection;
  * length of hospitalization;
  * rate of intraprocedural perforation;
  * rate of intraprocedural bleeding.
delayed perforation | at 1 months
  To compare the proportion of delayed perforation between the two groups
proportion of post-electrocoagulation syndrome | at Day 7
  To compare the proportion of post-electrocoagulation syndrome between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Humanitas Research Hospital, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Koyama Y, Fukuzawa M, Aikawa H, Nemoto D, Muramatsu T, Matsumoto T, Uchida K, Madarame A, Morise T, Yamaguchi H, Kono S, Nagata N, Sugimoto M, Kawai T, Saito Y, Itoi T. Underwater endoscopic submucosal dissection for colorectal tumors decreases the incidence of post-electrocoagulation syndrome. J Gastroenterol Hepatol. 2023 Sep;38(9):1566-1575. doi: 10.1111/jgh.16259. Epub 2023 Jun 15. PMID 37321649
- [Background] Yamamoto H, Hayashi Y, Despott EJ. The pocket-creation method for endoscopic submucosal dissection combined with saline-immersion: another potential option to overcome challenges in colorectal endoscopic submucosal dissection. Gastrointest Endosc. 2019 Aug;90(2):288-289. doi: 10.1016/j.gie.2019.04.244. No abstract available. PMID 31327340
- [Background] Capogreco A, Hassan C, De Blasio F, Massimi D, de Sire R, Galtieri PA, Despott EJ, Alkandari A, Bhandari P, Facciorusso A, Maselli R, Repici A. Prophylactic underwater vessel coagulation for submucosal endoscopy. Gut. 2024 Jun 6;73(7):1049-1051. doi: 10.1136/gutjnl-2024-332002. No abstract available. PMID 38383144
- [Background] Despott EJ, Hirayama Y, Lazaridis N, Koukias N, Telese A, Hayashi Y, Miura Y, Yamamoto H, Murino A. Saline immersion therapeutic endoscopy facilitated pocket-creation method for endoscopic submucosal dissection (with video). Gastrointest Endosc. 2019 Mar;89(3):652-653. doi: 10.1016/j.gie.2018.10.005. No abstract available. PMID 30784510
- [Background] Spadaccini M, Fuccio L, Lamonaca L, Frazzoni L, Maselli R, Di Leo M, Galtieri PA, Craviotto V, D'Amico F, Hassan C, Repici A. Underwater EMR for colorectal lesions: a systematic review with meta-analysis (with video). Gastrointest Endosc. 2019 Jun;89(6):1109-1116.e4. doi: 10.1016/j.gie.2018.10.023. Epub 2018 Oct 25. PMID 30862352
- [Background] Tseng CW, Hsieh YH, Lin CC, Koo M, Leung FW. Heat sink effect of underwater polypectomy in a porcine colon model. BMC Gastroenterol. 2021 Oct 27;21(1):406. doi: 10.1186/s12876-021-01985-1. PMID 34706664
- [Background] Lenz L, Martins B, Andrade de Paulo G, Kawaguti FS, Baba ER, Uemura RS, Gusmon CC, Geiger SN, Moura RN, Pennacchi C, Simas de Lima M, Safatle-Ribeiro AV, Hashimoto CL, Ribeiro U, Maluf-Filho F. Underwater versus conventional EMR for nonpedunculated colorectal lesions: a randomized clinical trial. Gastrointest Endosc. 2023 Mar;97(3):549-558. doi: 10.1016/j.gie.2022.10.033. Epub 2022 Oct 26. PMID 36309072
- [Background] Nagl S, Ebigbo A, Goelder SK, Roemmele C, Neuhaus L, Weber T, Braun G, Probst A, Schnoy E, Kafel AJ, Muzalyova A, Messmann H. Underwater vs Conventional Endoscopic Mucosal Resection of Large Sessile or Flat Colorectal Polyps: A Prospective Randomized Controlled Trial. Gastroenterology. 2021 Nov;161(5):1460-1474.e1. doi: 10.1053/j.gastro.2021.07.044. Epub 2021 Aug 8. PMID 34371000
- [Background] Binmoeller KF, Weilert F, Shah J, Bhat Y, Kane S. "Underwater" EMR without submucosal injection for large sessile colorectal polyps (with video). Gastrointest Endosc. 2012 May;75(5):1086-91. doi: 10.1016/j.gie.2011.12.022. Epub 2012 Feb 25. PMID 22365184
- [Background] Arezzo A, Passera R, Marchese N, Galloro G, Manta R, Cirocchi R. Systematic review and meta-analysis of endoscopic submucosal dissection vs endoscopic mucosal resection for colorectal lesions. United European Gastroenterol J. 2016 Feb;4(1):18-29. doi: 10.1177/2050640615585470. Epub 2015 May 5. PMID 26966519
- [Background] Stephane S, Timothee W, Jeremie A, Raphael O, Martin D, Emmanuelle P, Elodie L, Quentin D, Nikki C, Sonia B, Hugo L, Guillaume G, Romain L, Mathieu P, Sophie G, Jeremie J. Endoscopic submucosal dissection or piecemeal endoscopic mucosal resection for large superficial colorectal lesions: A cost effectiveness study. Clin Res Hepatol Gastroenterol. 2022 Jun-Jul;46(6):101969. doi: 10.1016/j.clinre.2022.101969. Epub 2022 Jun 1. PMID 35659602
- [Background] Jacques J, Schaefer M, Wallenhorst T, Rosch T, Lepilliez V, Chaussade S, Rivory J, Legros R, Chevaux JB, Leblanc S, Rostain F, Barret M, Albouys J, Belle A, Labrunie A, Preux PM, Lepetit H, Dahan M, Ponchon T, Crepin S, Marais L, Magne J, Pioche M. Endoscopic En Bloc Versus Piecemeal Resection of Large Nonpedunculated Colonic Adenomas : A Randomized Comparative Trial. Ann Intern Med. 2024 Jan;177(1):29-38. doi: 10.7326/M23-1812. Epub 2023 Dec 12. PMID 38079634
- [Background] Nishihara R, Wu K, Lochhead P, Morikawa T, Liao X, Qian ZR, Inamura K, Kim SA, Kuchiba A, Yamauchi M, Imamura Y, Willett WC, Rosner BA, Fuchs CS, Giovannucci E, Ogino S, Chan AT. Long-term colorectal-cancer incidence and mortality after lower endoscopy. N Engl J Med. 2013 Sep 19;369(12):1095-105. doi: 10.1056/NEJMoa1301969. PMID 24047059
- [Background] Schoen RE, Pinsky PF, Weissfeld JL, Yokochi LA, Church T, Laiyemo AO, Bresalier R, Andriole GL, Buys SS, Crawford ED, Fouad MN, Isaacs C, Johnson CC, Reding DJ, O'Brien B, Carrick DM, Wright P, Riley TL, Purdue MP, Izmirlian G, Kramer BS, Miller AB, Gohagan JK, Prorok PC, Berg CD; PLCO Project Team. Colorectal-cancer incidence and mortality with screening flexible sigmoidoscopy. N Engl J Med. 2012 Jun 21;366(25):2345-57. doi: 10.1056/NEJMoa1114635. Epub 2012 May 21. PMID 22612596
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2018. CA Cancer J Clin. 2018 Jan;68(1):7-30. doi: 10.3322/caac.21442. Epub 2018 Jan 4. PMID 29313949
- [Background] Arnold M, Sierra MS, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global patterns and trends in colorectal cancer incidence and mortality. Gut. 2017 Apr;66(4):683-691. doi: 10.1136/gutjnl-2015-310912. Epub 2016 Jan 27. PMID 26818619
- [Background] Morgan E, Arnold M, Gini A, Lorenzoni V, Cabasag CJ, Laversanne M, Vignat J, Ferlay J, Murphy N, Bray F. Global burden of colorectal cancer in 2020 and 2040: incidence and mortality estimates from GLOBOCAN. Gut. 2023 Feb;72(2):338-344. doi: 10.1136/gutjnl-2022-327736. Epub 2022 Sep 8. PMID 36604116